CLINICAL TRIAL: NCT05230966
Title: Immunometabolic Pattern of Intermittent Hypoxia as a Protective Mechanism Against Lethal Reperfusion Injury in Patients With ST-segment Elevation Myocardial Infarction
Brief Title: Immunometabolic Pattern of Intermittent Hypoxia During ST-segment Elevation Myocardial Infarction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Clinical Hospital Center Rijeka (Other)
Responsible Party: Principal Investigator, Koraljka Benko, M.D., Clinical Hospital Center Rijeka
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 2170-29-02/1-21-2
Record Dates: First submitted 2022-01-12; First posted 2022-02-09 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-01

CONDITIONS: Myocardial Ischemic-reperfusion Injury
MeSH Terms: conditions — Myocardial Reperfusion Injury

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Group 1- angina pectoris (No Intervention): Patients with acute coronary syndrome; angina pectoris (chest pain with negative troponin T with or without changes in electrocardiographic findings);
- Group 2 - angina pectoris + STEMI+ PCI (No Intervention): Patients with acute myocardial infarction with ST-segment elevation, < 6 hours from the onset of chest pain and preceding symptoms of angina pectoris with primary percutaneous coronary intervention.
- Group 3 - without angina pectoris + STEMi + RIC + PCI (Active Comparator): Patients with acute myocardial infarction with ST-segment elevation, < 6 hours from the onset of chest pain and without preceding symptoms of angina pectoris with primary percutaneous coronary intervention during which it's carried out remote ischemic conditioning (RIC)
  Interventions: Device: Remote Ischemic Conditioning (RIC)
- Group 4 - without angina pectoris + STEMI + PCI (No Intervention): Patients with acute myocardial infarction with ST-segment elevation, < 6 hours from the onset of chest pain and without preceding symptoms of angina pectoris with primary percutaneous coronary intervention.
- Group 5 - healthy + RIC (Active Comparator): healthy volunteers of the same age and sex, whose samples will be taken after the RIC procedure
  Interventions: Device: Remote Ischemic Conditioning (RIC)

INTERVENTIONS:
Device: Remote Ischemic Conditioning (RIC) — RIC is a non-invasive method that achieves a state of intermittent hypoxia, and is performed by inflating the cuff of the pressure gauge on the left upper arm to 200 mmHg in 4 episodes of five-minute ischemia and reperfusion alternately for 45 minutes.
  Arms: Group 3 - without angina pectoris + STEMi + RIC + PCI; Group 5 - healthy + RIC

SUMMARY:
The aim of this study is to characterize the protective pattern of intermittent hypoxia, angina pectoris and remote ischemic conditioning, in reperfusion injury by determining and monitoring the plasma immunometabolic parameters of patients with STEMI. This could contribute to better understanding of this phenotypic pattern with translation into clinical practice.

DETAILED DESCRIPTION:
In acute myocardial infarction with ST segment elevation (STEMI), lethal reperfusion injury of the myocardium, caused by percutaneous coronary intervention (PCI), represents additional and irreversible damage due to ischemic heart muscle reperfusion that contributes to the final size of the infarct zone by up to 50%. The size of the infarcted area is the major determinant for the long-term prognosis and heart failure progression in patients with STEMI. Cardioprotection from ischemic - reperfusion myocardial injury (MIRI) can be regulated by its own innate physiological adaptive mechanisms like intermittent hypoxia achieved by the method of conditioning that includes short sublethal ischemic and reperfusion episodes.

The known natural clinical equivalent of intermittent hypoxia and the starting point in understanding the underlying mechanism is angina pectoris (AP).

Intermittent hypoxia is a protective mechanism against heart ischemic-reperfusion injury with reduced tissue damage and consequently better outcome in patients with STEMI. For the purpose of this work, a cardioprotective pattern was defined that includes immunometabolic factors as parameters for assessing the state of intermittent hypoxia on which the success of the application of the method of remote ischemic conditioning (RIC) is based.

ELIGIBILITY:
Inclusion Criteria:

For group 1:

1. Acute coronary syndrome; angina pectoris (chest pain with negative troponin T with or without changes in electrocardiographic findings);
2. Monovascular disease, preocclusive stenosis with TIMI(thrombolysis in myocardial infarction) > 1 on the left main or anterior descending branch of the left coronary artery
3. Visually estimated diameter of the epicardial coronary artery from 2.5 mm to 4.0 mm

For group 2:

1. Acute myocardial infarction with ST-segment elevation (ST-segment elevation> 0.1 mV in two or more leads, or> 0.2 mV in V1-V3) <6 hours from the onset of chest pain
2. Symptoms of angina pectoris preceding acute myocardial infarction
3. Monovascular disease, occlusion or preocclusive stenosis of the anterior descending branch of the left coronary artery with TIMI <1 flow in STEMI;
4. After opening the artery and setting the stent TIMI> 2 flow
5. Visually estimated epicardial coronary artery diameter up to 2.5 mm to 4.0 mm

For groups 3 and 4:

1. Acute myocardial infarction with ST-segment elevation (ST-segment elevation> 0.1 mV in two or more leads, or> 0.2 mV in V1-V3) <6 hours from the onset of chest pain
2. No symptoms of angina pectoris preceding acute myocardial infarction
3. Monovascular disease, occlusion or preocclusive stenosis of the anterior descending branch of the left coronary artery with TIMI <1 flow in STEMI;
4. After opening the artery and stent placement TIMI> 2 flow
5. Visually estimated diameter of the epicardial coronary artery from 2.5 mm to 4.0 mm

For all groups:

1. Age of patients over 18 years
2. Signed written informed consent to be included in the survey

Exclusion Criteria:

1. Cardiac arrest before or after PCI;
2. Cardiogenic shock;
3. Previous myocardial infarction or revascularization of the heart;
4. Anginal pain before the onset of STEMI in patients to be subjected to RIC;
5. Patients with end-stage renal or hepatic disease, diabetics with developed micro and macrovascular complications, oncology patients;
6. Significant collaterals in the area of the occluded artery (Rentrop gradus> 1);
7. Previous use of nitrates and corticosteroids;
8. Pregnant or breastfeeding women;
9. Iodine allergy (contrast media);
10. Increase in body temperature > 37.5 ° C
11. Participation in another clinical trial

Randomly selected (coin toss) patients will be randomized to group 3 and 4, respectively, for percutaneous coronary intervention with or without RIC

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2022-02-01 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-03-02 (Estimated)

PRIMARY OUTCOMES:
Measurement of the concentration and dynamics of troponin T (Trop T) | 24 hour
  Serum concentrations (ng/ml) will be measured at four time points 0. - after coronary angiography and before PCI; 1. - 1 hour after PCI; 2. - 12 hours after PCI and 3. - 24 hours after PCI.
Measurement of the concentration and dynamics of cardiac myosin binding protein C (cMyBP-C) | 24 hour
  Serum concentrations (ng/ml) will be measured at four time points 0. - after coronary angiography and before PCI; 1. - 1 hour after PCI; 2. - 12 hours after PCI and 3. - 24 hours after PCI.
Measurement of the concentration and dynamics of creatine kinase-MB (CK-MB) | 24 hour
  Serum concentrations (ng/ml) will be measured at four time points 0. - after coronary angiography and before PCI; 1. - 1 hour after PCI; 2. - 12 hours after PCI and 3. - 24 hours after PCI.
Measurement of the concentration and dynamics of oxidation/mitochondrial parameter, hypoxia-induced factor 1 alpha (HIF 1α) | 24 hour
  serum concentrations (pg/ml) will be measured at four time points 0. - after coronary angiography and before PCI; 1. - 1 hour after PCI; 2. - 12 hours after PCI and 3. - 24 hours after PCI.
Measurement of the concentration and dynamics of metabolic parameter, glycine | 24 hour
  Serum concentrations (μmol/l) will be measured at four time points 0. - after coronary angiography and before PCI; 1. - 1 hour after PCI; 2. - 12 hours after PCI and 3. - 24 hours after PCI.
Measurement of the concentration and dynamics of metabolic parameter, kynurenine | 24 hour
  Serum concentrations (μmol/l) will be measured at four time points 0. - after coronary angiography and before PCI; 1. - 1 hour after PCI; 2. - 12 hours after PCI and 3. - 24 hours after PCI.
Measurement of the concentration and dynamics of metabolic parameter, succinate | 24 hour
  Serum concentrations (μM) will be measured at four time points 0. - after coronary angiography and before PCI; 1. - 1 hour after PCI; 2. - 12 hours after PCI and 3. - 24 hours after PCI.
Measurement of the concentration and dynamics of immunological parameter, interleukin 1 beta (IL-1 beta) | 24 hour
  Serum concentrations (pg/ml) will be measured at four time points 0. - after coronary angiography and before PCI; 1. - 1 hour after PCI; 2. - 12 hours after PCI and 3. - 24 hours after PCI.
Measurement of the concentration and dynamics of immunological parameter, transforming growth factor beta (TGF beta) | 24 hour
  Serum concentrations (ng/ml) will be measured at four time points 0. - after coronary angiography and before PCI; 1. - 1 hour after PCI; 2. - 12 hours after PCI and 3. - 24 hours after PCI.
Measurement of the concentration and dynamics of immunological parameter, monocyte chemoattraction protein 1 (MCP-1) | 24 hour
  Serum concentrations (pg/ml) will be measured at four time points 0. - after coronary angiography and before PCI; 1. - 1 hour after PCI; 2. - 12 hours after PCI and 3. - 24 hours after PCI.

SECONDARY OUTCOMES:
The changes in serum values of immunometabolic parameters and creatine kinase-MB | 24 hour
  The data of immunometabolic parameters at baseline and during follow up period (measured at 0, 1, 12 and 24 hours after the intervention) in three groups of patients with PCI will be compared with a degree of tissue damage creatine kinase-MB.
The changes in serum values of immunometabolic parameters and troponin T | 24 hour
  The data of immunometabolic parameters at baseline and during follow up period (measured at 0, 1, 12 and 24 hours after the intervention) in three groups of patients with PCI will be compared with a degree of tissue damage troponin T
The changes in serum values of immunometabolic parameters and left heart ejection fraction | 7 day
  The data of immunometabolic parameters at baseline and during follow up period (measured at 0, 1, 12 and 24 hours after the intervention) in three groups of patients with PCI will be compared with functional assessment of the heart muscle, ejection fraction (%).
The changes in serum values of immunometabolic parameters in PCI groups and angina pectoris (AP) group | 24 hour
  The data of immunometabolic parameters at baseline and during follow up period (measured at 0, 1, 12 and 24 hours after the intervention) in three groups of patients with PCI will be compared with the data of patients diagnosed with angina pectoris (AP).
The changes in serum values of immunometabolic parameters in PCI groups and the group of healthy volunteers | 24 hour
  The data of immunometabolic parameters at baseline and during follow up period (measured at 0, 1, 12 and 24 hours after the intervention) in three groups of patients with PCI will be compared with the group of healthy volunteers in whom the RIC method was used.

CONTACTS AND LOCATIONS:
Overall Officials: Koraljka Benko, MD, Principal Investigator — CHC Rijeka; Croatia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hausenloy DJ, Yellon DM. Myocardial ischemia-reperfusion injury: a neglected therapeutic target. J Clin Invest. 2013 Jan;123(1):92-100. doi: 10.1172/JCI62874. Epub 2013 Jan 2. PMID 23281415
- [Background] Hausenloy DJ. Cardioprotection techniques: preconditioning, postconditioning and remote conditioning (basic science). Curr Pharm Des. 2013;19(25):4544-63. doi: 10.2174/1381612811319250004. PMID 23270554
- [Background] Han X, Jeong MH, Won J, Kim Y, Kim MC, Sim DS, Hong YJ, Kim JH, Ahn Y. Impact of Previous Angina on Clinical Outcomes in ST-Elevation Myocardial Infarction Underwent Percutaneous Coronary Intervention. Chonnam Med J. 2020 May;56(2):136-143. doi: 10.4068/cmj.2020.56.2.136. Epub 2020 May 25. PMID 32509561
- [Background] Heusch G, Botker HE, Przyklenk K, Redington A, Yellon D. Remote ischemic conditioning. J Am Coll Cardiol. 2015 Jan 20;65(2):177-95. doi: 10.1016/j.jacc.2014.10.031. PMID 25593060